CLINICAL TRIAL: NCT05584163
Title: Single-center, Randomized, Prospective Controlled Pilot Study to Evaluate the Prevention and Safety of Doxorubicin-induced Cardiomyopathy Using Extracorporeal Shock Waves in Breast Cancer Patients Using Doxorubicin Anticancer Drugs
Brief Title: Pilot Study to Evaluate the Prevention and Safety of Doxorubicin-induced Cardiomyopathy Using Extracorporeal Shock Waves
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Ewha Womans University Mokdong Hospital (Other)
Responsible Party: Principal Investigator, Kihwan Kwon, Professor, Ewha Womans University Mokdong Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 2020-12-044-012
Record Dates: First submitted 2022-10-12; First posted 2022-10-18 (Actual); Last update posted 2023-06-02 (Actual); Status verified 2023-05

CONDITIONS: Breast Cancer
Keywords: Chemotherapy induced cardiomyopathy
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control group (No Intervention): Group not using drugs used for the prevention of cardiomyopathy caused by doxorubicin, including extracorporeal shock wave
- ESWT treatment group (Experimental): Group receiving extracorporeal shock wave therapy
  Interventions: Device: Extracorporeal shock waves

INTERVENTIONS:
Device: Extracorporeal shock waves — 3 times of extracorporeal shock wave therapy is performed, and 1 cycle of extracorporeal shock wave therapy is performed (every 6 weeks) every 2 cycles of chemotherapy. Echocardiography is performed at baseline and every 4 cycles of chemotherapy.
  Arms: ESWT treatment group

SUMMARY:
Until now, patients receiving doxorubicin chemotherapy should use only the cumulative dose related to known cardiotoxicity, or if cardiotoxicity occurs below the known cumulative dose, use of doxorubicin as chemotherapy should be stopped. In this study, in patients with normal heart function receiving doxorubicin chemotherapy, extracorporeal shock wave therapy was performed 3 times a week during chemotherapy, and 1 cycle of extracorporeal shock wave therapy was performed (every 6 weeks) every 2 cycles of chemotherapy. Echocardiography should be performed at baseline and every 4 cycles of chemotherapy, and follow-up 3 months after chemotherapy is completed to compare the incidence of cardiomyopathy caused by chemotherapy between the two groups.

DETAILED DESCRIPTION:
1. Extracorporeal shock wave therapy cycle

   * For breast cancer patients using doxorubicin as the main anticancer agent, 1 cycle of extracorporeal shock wave therapy was performed every 2 cycles of chemotherapy.
   * The extracorporeal shock wave therapy is targeted to the existing refractory angina pectoris patients and is based on the energy used in patients with ischemic heart disease without serious side effects. The treatment is performed 3 times a week in 1 cycle, 200 shots per spot. , a shock wave of 0.09mJ/mm2 energy was applied to 40-60 spots (8,19,20)
   * Conventional chemotherapy is performed every 3 weeks, and the dose of doxorubicin used per session is 40-60 mg/m2, and considering the cumulative dose, chemotherapy is performed on average 6-8 times. Therefore, extracorporeal shock wave therapy is performed every 6 weeks, and a total of 3 to 4 times.
   * It is expected that factors affecting efficacy will be controlled by targeting patients with the same carcinoma, the same chemotherapy, and no underlying heart disease. Since the cumulative doxorubicin dose can be received from a minimum of 60mg/m2 to a maximum of 400mg/m2, the cumulative dose of doxorubicin in the control and experimental groups should be divided into sections to further analyze the cardiomyopathy incidence rate and echocardiographic indicators.
   * Extracorporeal shock wave therapy position and posture The extracorporeal shock wave probe is placed at the position where the apical view of the echocardiogram is taken, and the patient's posture is supine or lateral position. When extracorporeal shock wave therapy is performed in the following locations, the entire cardiac muscle can be included.
2. It was assumed that the incidence of cardiomyopathy in patients receiving extracorporeal shock wave therapy was low. Cardiomyopathy is defined as ① a decrease in the absolute value of left ventricular ejection fraction by 10% or more or ② a decrease in the absolute value of LV global longitudinal strain (GLS) by 8% or more. In this study, cardiomyopathy caused by the definition of LV global longitudinal strain (GLS) was set as the primary efficacy evaluation.

   Therefore, when the target number of subjects is set according to the definition that the LV global longitudinal strain (GLS) set as the primary efficacy evaluation variable is reduced to less than 17.5%, the absolute LVGLS value is the dependent variable, the significance level is 0.05, and the power is based on 85%. Therefore, when the ratio between groups is 1:1, the mean of the treated group is expected to be 19.6%, the mean of the untreated group is expected to be 18.0%, and when the standard deviations are applied as 2.4% and 2.4%, respectively, when using the G*Power 3.1 program, 33 people are required for each calculated group. Considering the dropout rate of 10%, 36 people each, a total of 72 subjects, is calculated as the required number of subjects.
3. Observational items/clinical examination items and observational examination method Basic information: Acquired at the time of clinical research registration

   * Age, gender, height, weight, BMI, systolic diastolic blood pressure, pulse clinical information
   * Clinical information 1: Acquired at the time of clinical research registration Accompanying diseases (hypertension, diabetes, dyslipidemia, chronic kidney disease, etc.), past acute reaction
   * Clinical information 2: Acquired at the time of clinical study registration and every echocardiogram follow-up Breast cancer stage, doxorubicin dose used for chemotherapy, chemotherapy cycle medications taken within the past 4 weeks (including current medications);
   * Diagnostic test results (Creatinie Kinase (CK), Creatine Kinase-MB (CK-MB), Troponin T (TnT), N-terminal pro-Brain natriuretic peptide (NT-proBNP), compete blood count (CBC), Chemistry) ,
   * New York Heart Association (NYHA) classiciation - Class 1,2,3,4; It is obtained by dividing into Class 1, 2, 3, and 4 through a questionnaire about the patient's subjective symptoms, and is obtained through a questionnaire at the time of clinical study registration and every echocardiogram follow-up.
   * Electrocardiogram (EKG). Chest X-ray (CXR) Echocardiographic parameters: Acquired at the time of clinical study registration and at each echocardiographic follow-up.

Left ventricular ejection fraction (LVEF), Left ventricular end-diastolic dimension (LVEDD), Left ventricular end-systolic dimension (LVESD), Inter-ventricular septal diastolic phase (IVSd), Posterior wall thickness (PWd), Mitral inflow pattern, Mitral valve tissue doppler, Rightly ventricular systolic pressure (RVSP), Left ventricular (LV) global longitudinal strain

ELIGIBILITY:
Inclusion Criteria:

1. Breast cancer patients receiving doxorubicin chemotherapy (for patients with operable breast cancer who receive doxorubicin with neoadjuvant or adjuvant chemotherapy)
2. Patients who are expected to receive at least 3 cycles of doxorubicin chemotherapy after registration and who can receive at least 2 extracorporeal shock wave therapy
3. Those with a left ventricular ejection fraction of 50% or more at screening

Exclusion Criteria:

1. Subjects under the age of 19
2. Those who have implanted an intracardiac device (implantable defibrillator, pacemaker)
3. Hemodynamically unstable ventricular tachycardia confirmed
4. If you have QT prolongation syndrome or are receiving medication that increases QT interval

   * Antiarrhythmics class IA; quinidine, procainamide
   * Antiarrhythmics class III; amiodarone, sotalol
5. Patients with atrial fibrillation or those who have undergone defibrillation for atrial fibrillation within the last 3 months
6. In case of structural heart disease (congenital heart disease, valvular disease, etc.) and related surgery
7. Persons who have had coronary artery disease or a subsequent PCI or coronary artery bypass surgery
8. Those with symptoms of unstable angina requiring hospitalization
9. Persons suspected or diagnosed with cardiomyopathy due to causes other than chemotherapy
10. When life expectancy is less than 6 months
11. Pregnant women or those planning to become pregnant
12. Moderate or severe hepatic impairment (ex. Child-Pugh class B,C)
13. Creatinine clearance < 30mL/min
14. Patients judged to be inappropriate by other researchers

Min Age: 19 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 72 (Estimated)
Dates: Start 2020-10-01 (Actual); Primary Completion 2023-06 (Estimated); Study Completion 2023-06 (Estimated)

PRIMARY OUTCOMES:
Chemotherapy induced cardiomyopathy | 3months, 6months
  Primary efficacy endpoint: Cardiomyopathy is defined as the LV longitudinal strain value, an echocardiographic index, and the incidence rate of cardiomyopathy between the experimental group and the control group is compared. The definition of cardiomyopathy in LV longitudinal strain is as follows
  - When the strain value of the longitudinal axis of the left ventricle (LV global longitudinal strain) decreases to less than -17.5% or reduction of >15% compared to the baseline value.

SECONDARY OUTCOMES:
Chemotherapy induced cardiomyopathy 2 | 3months, 6months
  Secondary efficacy endpoint: To compare the rate of cardiomyopathy between the experimental group and the control group in breast cancer patients receiving doxorubicin-containing chemotherapy with baseline normal heart function. The definition of cardiomyopathy is as follows.
  * A decrease of more than 10% in absolute left ventricular ejection fraction (LVEF) or
  * A decrease of less than 50% from the normal range of left ventricular ejection fraction (>55%)

CONTACTS AND LOCATIONS:
Overall Officials: Shinjeong Song, MD, Study Director — EUMC
Locations (1):
- Kiwhan Kim, Seoul, Yangcheon Gu, South Korea

IPD SHARING:
Plan to Share IPD: No
IPD are not to be shared with other researchers.

REFERENCES:
- [Derived] Song S, Woo J, Kim H, Lee JW, Lim W, Moon BI, Kwon K. A prospective randomized controlled trial to determine the safety and efficacy of extracorporeal shock waves therapy for primary prevention of subclinical cardiotoxicity in breast cancer patients without a cardiovascular risk treated with doxorubicin. Front Cardiovasc Med. 2024 Feb 7;11:1324203. doi: 10.3389/fcvm.2024.1324203. eCollection 2024. PMID 38385137
- See also: Extracorporeal shock waves protect cardiomyocytes from doxorubicin-induced cardiomyopathy by upregulating survivin via the integrin-ILK-Akt-Sp1/p53 axis — https://www.nature.com/articles/s41598-019-48470-0